CLINICAL TRIAL: NCT04960527
Title: The Acute Effects of Tart Cherry Juice on Uric Acid and Biomarkers of Cardiovascular Disease Risk in Healthy Individuals
Brief Title: Acute Effects of Tart Cherry on Uric Acid and Biomarkers of CVD Risk in Healthy Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Hallam University (Other)
Responsible Party: Principal Investigator, Tony Lynn, Principal Lecturer Ethics Lead, Sheffield Hallam University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: ER9199256
Record Dates: First submitted 2021-07-02; First posted 2021-07-14 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Uric Acid; Cardiovascular Diseases; Gout
MeSH Terms: conditions — Cardiovascular Diseases; Gout | interventions — Water

STUDY DESIGN:
Intervention Model Description: 2-way crossover, randomised controlled trial. Participants will be allocated to consume tart cherry juice or a neutral water control on separate occasions. The order of this allocation will be randomised.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tart cherry juice (Experimental): 30 mL tart cherry concentrate (CherryActive, UK, 100% Montmorency) diluted with 220 mL water (totalling 250 mL). According to available manufacturers data, this is equivalent to consuming 90-100 fresh cherries.
  Interventions: Dietary Supplement: Tart cherry juice
- Water (Other): 250 mL water (neutral control)
  Interventions: Other: Water

INTERVENTIONS:
Dietary Supplement: Tart cherry juice — 250 mL tart cherry juice (30 mL tart cherry concentrate [CherryActive, UK] diluted with 220 mL water) is consumed on a single occasion by each participant. This will be consumed immediately following the baseline measurements one laboratory visit.
  Arms: Tart cherry juice
Other: Water — 250 mL water is consumed on a single occasion by each participant. This will be consumed immediately following the baseline measurements one laboratory visit.
  Arms: Water

SUMMARY:
This study aims to provide evidence as to whether consumption of tart cherry juice can reduce the risk of gout and cardiovascular disease (CVD) in an acute context. The proposed study is a 2-way cross-over, randomised, placebo-controlled trial and aims to answer the following research questions:

1. What effect does a single 30mL serving of tart cherry concentrate have on serum uric acid and urinary excretion of uric acid in healthy individuals, when compared with water?
2. What effect does a single 30mL serving of tart cherry concentrate have on markers of cardiovascular disease risk and oxidative stress in healthy individuals, when compared with water?

By measuring acute changes in serum urate, fractional urinary urate excretion, inflammatory markers, oxidative stress markers and CVD risk markers (namely central and brachial blood pressure, and arterial stiffness), it will highlight possible mechanisms through which tart cherry may reduce risk of gout and/or CVD.

DETAILED DESCRIPTION:
Healthy, non-smoking, adult volunteers (n = 15) will be recruited to a 2-way cross-over, randomized, placebo-controlled study.

A sample size of 13 has been calculated using data from White et al. (2018), using the primary outcome of change in serum uric acid level. Between-person variations in serum urate was established at approximately 50 µmol/L. Within-subject variation to apple juice was approximately 35 µmol/L. It has been estimated that cherry juice will produce a fall in serum urate of approximately 15 µmol/L (Jacob et al., 2003). Therefore, 13 participants will be needed to detect this change with 80% power at an alpha level of 0.05.

Participants will avoid strenuous exercise for 72-hours prior to the study until 24-hours post-consumption of the test drinks; compliance will be assessed through completion of a physical activity diary. They will also follow a low-polyphenolic diet for 48-hours prior to the study until 24-hours post-consumption of the test drinks; participants will be provided with a list of foods/drinks to avoid and compliance will be assessed through completion of a food diary. Participants will be provided with instructions of foods to avoid and a low polyphenolic pasta ready-meal, dessert and low nitrate water to consume the evening preceding the study day.

Participants will attend the laboratory following an overnight fast. Blood pressure (central and brachial) and arterial stiffness will be measured using a non-invasive Vicorder device. A venepuncture blood sample will be collected by a researcher trained in phlebotomy before consumption of the test drink. Approximately 10 ml of blood will be taken during each venepuncture. A urine sample will also be collected. Participants will consume 250 ml of tart cherry juice or neutral control (water) on two occasions, at least one week apart; the sequence order will be random. The cherry juice comprises 30 mL tart cherry concentrate diluted with 220 mL water. Further venous blood samples will be taken at 1 and 2 hours post-consumption. These will be supplemented with finger-prick samples collected at 3, 5 and 24 hours post drink. Post-drink measures of arterial stiffness will be taken at 1, 2, 3, 5 and 24-hours post-consumption. Additional urine samples will also be collected between 0-2, 2-4, 4-5, 5-8, 8-11, and 11-24 hours, post-consumption of the test drinks. Participants' water intake during each laboratory visit will be standardised at 500 ml. Participants will be provided with a low-polyphenolic sandwich lunch, pasta ready-meal dinner, dessert, snacks and low nitrate water to consume following the 5-hour measurements. Participants will return to the laboratory the next morning following a 12-hour fast for their 24-hour measurements.

Blood will be analysed for serum uric acid and creatinine concentrations at all time points and for CRP (a measure of inflammation) at baseline, 2, and 5 hours, post-drink. White blood cells (lymphocytes) will be separated from whole venous blood samples collected at baseline, 1 and 2-hours post-drink consumption for the analysis of oxidative DNA damage. Urine samples will be analysed for uric acid and creatinine to calculate fractional excretion of urinary uric acid (using a commercial colorimetric assay). Polyphenolic metabolites from the test drink will also be analysed in urine samples.

Data analysis: The effect of the treatment (tart cherry versus water) on all outcome variables will be analysed with 2-way repeated measures ANOVAs. A statistical significance level of P≤ 0.05 will be set.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or over
* able and willing to participate in the study and provide written informed consent

Exclusion Criteria:

* current smoker
* any known food allergies/intolerances
* history of medical conditions, including gastrointestinal disease, severe renal impairment (estimated glomerular filtration rate of <30ml/min) or renal disease, cardiovascular disease, diabetes (type 1 or type 2) and gout

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-07-10 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Change in serum urate (in millimoles per litre (mmol/l) | Measured at baseline, 1, 2, 3, 5 and 24 hours post-consumption of test drink
  Difference in serum urate in tart cherry juice arm versus water arm from baseline to 24 hours post-consumption of drink. Measured using a commercial fluorometric/colorimetric urate assay kit.

SECONDARY OUTCOMES:
Change in urinary urate (mmol/l) | Measured from samples collected at baseline and between 0-2 hours, 2-4 hours, 4-5 hours, 5-8 hours, 8-11 hours and 11-24 hours
  Difference in urinary urate in tart cherry juice arm versus water arm from baseline to 24 hours post-drink consumption. Measured using a commercial fluorometric/colorimetric assay kit
Change in urinary creatinine (mmol/l) | Measured from samples collected at baseline and between 0-2 hours, 2-4 hours, 4-5 hours, 5-8 hours, 8-11 hours and 11-24 hours
  Difference in urinary creatinine in tart cherry juice arm versus water arm from baseline hours to 24 hours post-drink consumption. Measured using a commercial fluorometric/colorimetric assay kit
Change in serum creatinine (mmol/l) | Measured at baseline, 1, 2, 3, 5 and 24 hours post-consumption of test drink
  Difference in serum creatinine in tart cherry juice arm versus water arm from baseline to 24 hours post-drink consumption. Measured using a commercial fluorometric/colorimetric assay kit
Change in c reactive protein (in milligrams per litre (mg/l) | Measured at baseline, 2 and 5 hours post-consumption of test drink
  Difference in serum c reactive protein (CRP) in tart cherry juice arm versus water arm from baseline to 5 hours post-consumption of drink. Measured using an enzyme-linked immunosorbent assay (ELISA).
Change in blood pressure (in millimetres of mercury (mmHg)) | Measured at baseline, 1, 2, 3, 5, and 24-hours post-consumption of test drink
  Difference in brachial and central blood pressure in tart cherry juice arm versus water arm from baseline to 24 hours post-consumption of drink. Measured using a Vicorder non-invasive device.
Change in arterial stiffness (Augmentation index measured in %, pulse wave velocity measured in meters per second (m/s)) | Measured at baseline, 1, 2, 3, 5, and 24-hours post-consumption of test drink
  Difference in augmentation index (AI) and pulse wave velocity (PWV) in tart cherry juice arm versus water arm from baseline to 24 hours post-consumption of drink. Measured using a Vicorder non-invasive device.
Change in oxidative damage (in percentage (%) of tail DNA) | Measured at baseline, 1 and 2 hours post-consumption of test drink
  Difference in markers of oxidative stress in tart cherry juice arm versus water arm from baseline to 2 hours post-consumption of drink. Measured using single-cell electrophoresis 'comet assay' as 8-oxo-dg levels in lymphocytes.

OTHER OUTCOMES:
Avoidance of strenuous physical activity | Measured from 72-hours prior to the study until 24-hours post-consumption of test drink
  Avoidance of strenuous exercise will be measured for 72-hours prior to the study until 24-hours post-consumption of both test drinks; compliance will be assessed through completion of a physical activity diary during this period.
Adherence to a low-polyphenolic diet | Measured from 48-hours prior to the study until 24-hours post-consumption of test drink
  Adherence to a low-polyphenolic diet for 48-hours prior to the study until 24-hours post-consumption of both test drinks (participants provided with a list of foods/drinks to avoid). Compliance assessed through completion of a food diary during this period.

CONTACTS AND LOCATIONS:
Overall Officials: Tony Lynn, PhD, Principal Investigator — Sheffield Hallam University
Locations (1):
- Food and Nutrition Group, Sheffield Hallam University, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jacob RA, Spinozzi GM, Simon VA, Kelley DS, Prior RL, Hess-Pierce B, Kader AA. Consumption of cherries lowers plasma urate in healthy women. J Nutr. 2003 Jun;133(6):1826-9. doi: 10.1093/jn/133.6.1826. PMID 12771324
- [Background] White SJ, Carran EL, Reynolds AN, Haszard JJ, Venn BJ. The effects of apples and apple juice on acute plasma uric acid concentration: a randomized controlled trial. Am J Clin Nutr. 2018 Feb 1;107(2):165-172. doi: 10.1093/ajcn/nqx059. PMID 29529161
- [Background] Lynn A, Mathew S, Moore CT, Russell J, Robinson E, Soumpasi V, Barker ME. Effect of a tart cherry juice supplement on arterial stiffness and inflammation in healthy adults: a randomised controlled trial. Plant Foods Hum Nutr. 2014 Jun;69(2):122-7. doi: 10.1007/s11130-014-0409-x. PMID 24570273
- [Background] Chai SC , Davis K , Wright RS , Kuczmarski MF , Zhang Z . Impact of tart cherry juice on systolic blood pressure and low-density lipoprotein cholesterol in older adults: a randomized controlled trial. Food Funct. 2018 Jun 20;9(6):3185-3194. doi: 10.1039/c8fo00468d. PMID 29862410
- [Background] Bell, P. G., Gaze, D. C., Davison, G. W., George, T. W., Scotter, M. J., & Howatson, G. (2014). Montmorency tart cherry (Prunus cerasus L.) concentrate lowers uric acid, independent of plasma cyanidin-3-O-glucosiderutinoside. Journal of Functional Foods, 11, 82-90.